CLINICAL TRIAL: NCT01543295
Title: Qualitative Evaluation of the DPP Syphilis Screen and Confirm Rapid Test to Detect the Presence of Antibodies Against Non-Treponemal and Treponema Pallidum Antigens in Fingerstick Whole Blood, Venous Whole Blood, Serum and Plasma Specimens.
Brief Title: Evaluation of the Performance of Chembio's DPP(R) Syphilis Screen & Confirm Rapid Test System
Status: Withdrawn | Type: Observational
Sponsor: Chembio Diagnostic Systems, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CP-SYP-01
Record Dates: First submitted 2011-08-08; First posted 2012-03-02 (Estimated); Last update posted 2015-07-29 (Estimated); Status verified 2015-07

CONDITIONS: Syphilis
Keywords: Non-Treponemal; Treponemal
MeSH Terms: conditions — Syphilis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Known Positive Syphilis Infection: Individuals known to have a clinical diagnosis of Syphilis
- High Risk for Syphilis Infection: Individuals with previous and confirmed STD infection, MSM, persons with high risk sexual behavior or clinical examination with classic manifestations of syphilis.
- Pregnant Women (High Risk and Low Risk): 1st or 3rd trimester from either High Risk (see description above) or Low Risk population.
  Low Risk are individuals not known to belong to any of the defined high-risk groups - i.e. "healthy patients" presenting for routine physicals or other unrelated non-life threatening illnesses, or individuals from a general low risk population such as students, employees of academic or other institutions, etc…

SUMMARY:
This study has been designed to evaluate the performance of the Chembio Diagnostics Systems, Inc. DPP® Syphilis Screen and Confirm rapid test. The device is intended to qualitatively and simultaneously detect the presence of antibodies to Non-treponemal and Treponema pallidum antigens in whole blood (capillary and venous), serum or plasma.

DETAILED DESCRIPTION:
Syphilis is a sexually transmitted disease (STD) caused by the spirochete Treponema pallidum. It is a chronic bacterial infection that remains a public health concern worldwide, especially in resource poor settings. Syphilis can be transmitted from infected women to their unborn children during pregnancy. Worldwide 12 million individuals are diagnosed with syphilis each year, 90% of them in developing countries. Diagnosed individuals are also at risk of becoming infected with and transmitting HIV [1].

Early and appropriate diagnosis and treatment prevents the transmission and development of severe complications. A rapid serologic test for specific antibodies to non-Treponemal and T. pallidum antigens is important in the early diagnosis and treatment monitoring of syphilis patients. In turn, this monitoring allows for the formulation of a more successful public health strategy. Various serologic tests are currently available such as Venereal Disease Research Laboratory (VDRL), rapid plasma reagin (RPR), fluorescent Treponemal antibody absorption (FTA-ABS) test, T. pallidum hemagglutination (TPHA) test, immunoenzymatic assay (EIA), Treponema pallidum particle agglutination (TPPA) test and Western blot (WB) test [2- 5]. The Chembio DPP Syphilis Screen & Confirm Assay is a unique non-Treponemal and Treponemal rapid point-of-care test, which is simple and easy to use. The DPP Syphilis Screen & Confirm Assay is a qualitative immunoassay for the detection of antibodies to the non-Treponemal and T. pallidum antigens in serum, plasma and whole blood.

ELIGIBILITY:
Inclusion Criteria:

* Must be at least 13 years of age (no upper age limit).
* Must be willing and able to receive post-test counseling, if applicable.
* Must sign (and be given) a copy of the written Informed Consent form and or Assent form (if applicable).
* Must be able to sustain fingersticks and venipuncture from the arm or hand only.

Exclusion Criteria:

* Persons who are under 13 years of age
* Persons who are unable to sustain venipuncture (as determined by investigator)
* Have previously participated in this clinical trial
* Persons who do not provide an informed consent, or withdraw consent.

Min Age: 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Participants will be recruited from study sites at diverse geographical locations in the United States. Such sites include primary care clinics, Obstetric/Gynecology clinics, physician offices, hospitals.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2011-07; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Clinical Performance Characteristics | 12 months
  Support the claims that the DPP Syphilis Screen and Confirm test system is:
  1. substantially equivalent to a recognized laboratory method for syphilis presumptive screening tests, and
  2. substantially equivalent to a recognized laboratory method for syphilis confirmatory tests.

SECONDARY OUTCOMES:
Specimen Types | 20 minutes
  The device detects specific antibodies to Non-Treponema and Treponema pallidum antigens in a variety of sample matrices: capillary whole blood, venous whole blood (with EDTA or heparin anticoagulant),serum and plasma (with EDTA or heparin anticoagulant).

CONTACTS AND LOCATIONS:
Overall Officials: Neil T Constantine, Ph.D, Principal Investigator — University of Maryland, Baltimore; Anthony LaMarca, M.D., Principal Investigator — Therafirst Medical Center; Neva Yeganeh, M.D., Principal Investigator — University of California, Los Angeles, David Geffen School of Medicine
Locations (3):
- United States (3):
  - Mattel Childrens Hospital, University of California, David Geffen School of Medicine, Los Angeles, California
  - Therafirst Medical Center, Fort Lauderdale, Florida
  - University of Maryland, Baltimore, Maryland